CLINICAL TRIAL: NCT05614856
Title: Aorto-iliac Occlusion Treatment With ShorT Unibody aorTic Endograft - ASTUTE Study
Acronym: ASTUTE
Status: Suspended | Type: Observational
Why Stopped: Local ethics committee concern
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Collaborators: Careggi Hospital (Other); Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other); Azienda Policlinico Umberto I (Other); S. Andrea Hospital (Other); Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Palermo (Other); Azienda USL Reggio Emilia - IRCCS (Other Government); Ospedale Policlinico San Martino (Other); Azienda Ospedaliero, Universitaria Pisana (Other); Azienda Ospedaliera Sant'Anna (Other)
Responsible Party: Principal Investigator, Roberto Silingardi, MD, Associate Professor in Vascular Surgery, Chief of department, Azienda Ospedaliero-Universitaria di Modena
Other Study IDs: ASTUTE
Record Dates: First submitted 2022-10-31; First posted 2022-11-14 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Occlusive Arterial Disease
Keywords: EVAR; AIOD; Unibody endograft
MeSH Terms: conditions — Arterial Occlusive Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Treatment Group: Patients affected by AIOD classified as TASC B, C or D involving aortic bifurcation and or the first 5mm of one of both common iliacs treated with the unibody endograft AFX (Endologix, Irvine, Calif)
  Interventions: Device: EVAR off-label use

INTERVENTIONS:
Device: EVAR off-label use — Normally a femoral access was used, although a brachial approach can be useful for crossing total occlusions. For TASC B and C lesions, predilatation of the iliac lesions is advisable, while for TASC D it is mandatory. In case of total aortic occlusions, the procedure demands that recanalization of the distal aorta occurs as close as possible to the bifurcation.. The key technique is to recanalize from one common iliac artery into the opposing snaring the wire to create a femoral-femoral crossover. The femoral-femoral wire is then replaced with a MPA catheter; the SurePass wire attached to the contralateral limb is then passed through the catheter. The sheath can be placed within 5 cm of the aortic bifurcation, and the AFX can be delivered through the common iliac and aortic occlusion. Predilatation were performed with bilateral 6-8 mm x 150 mm balloons and or progressive dilatators.
  Other Names: Aorto-iliac recanalization with an abdominal aortic endograft

SUMMARY:
The goal of this multi center prospective observational study is to evaluate the iliac patency rate during the time in patients treated with "AFX (Endologix, Irvine Calif)" unibody stent-graft for aorto-iliac occlusive disease The main question it aims to answer is if The Unibody AFX (Endologix) endograft could be in a large and real-world cohort of patients effective solution for the less-invasive treatment of the aortoiliac occlusive disease (AIOD).

Participants affected by AIOD with an indication of endovascular treatment will be prospectively enrolled and treated as our clinical practice. The requested follow-up did not differ from the one suggested by the most recent guidelines

DETAILED DESCRIPTION:
In the last two decades there was a general shift from conventional open surgery to endovascular mini-invasive interventions, particularly towards patients with iliac and aortic occlusive disease (AIOD). However, while iliac artery angioplasty and stenting increased 8.5 fold from 1996 to 2000, aorto-bifemoral bypass fell by only 15%1,2. Indeed, according to European Society of Vascular Surgery/European Society of cardiology guidelines, open surgery remains the preferred choice for the most complex lesions to address by in endovascular fashion (TransAtlantic Inter-Society Consensus [TASC II] type C and D lesions). The reason is the good long-term patency of aorto-bi-iliac or aorto-bifemoral bypass among endovascular devices. Surgery, however, is associated with a high burden of early and late morbidity and mortality, and this aggressive approach is limited by the patient's age and comorbidity. In 1991 the kissing stent technique emerged as an alternative for bilateral aortoiliac occlusive disease. Even if the reported technical success rates varied between 89% and 100% with a 1-year primary patency between 76% and 98%, outcomes may be worse in more complex lesions owing to radial size mismatch between stents and certain stent configurations within the distal aorta. In addition, heavy calcified or thrombus-filled aorta could increase technical complexity and risk of limb and life-threatening procedural complications such as dissections, aortic rupture, and peripherical embolizations. Covered stents may increase patency rates in extensive disease, as shown by The Covered vs Balloon Expandable Stent Trial (COBEST) and confirmed in various case series but did not address the problem of a potential radial size mismatch that can lead to re-circulation, turbulence, and stasis of blood, which in turn, may cause thrombus formation and intimal neohyperplasia. Another endovascular procedure for the treatment of AIOD is the CERAB technique. A CERAB is defined as an "endovascular reconstruction of the aortic bifurcation" using at least one covered stent-graft for the infrarenal aorta (flared proximally) and 2 stent-grafts deployed within the aortic stent and into the common iliac arteries. This particular configuration leads to the reduction of the radial mismatch, which is defined as the discrepancy between the stented lumen and the vessel lumen after stent placement and, as a result, to more favorable flow conditions. In addition, it protects against potentially fatal aortoiliac rupture during the dilatation of heavily calcified lesions. However, the radial mismatch is increased if the limbs are placed higher than the nonflared aortic stent. In addition, while the CERAB technique does recreate the aortic bifurcation, future crossover interventions may be more difficult. This is similar to most bifurcated aortic stent-grafts where the angle of engagement at the flow divider makes up-and-over access more challenging. Finally, dead space outside the proximal aortic stent can result in cases of aortic diameters > 20 mm. The aortic stent is then left protruding mal-opposed in a dilated aorta. Hence, this technique may not be indicated in the setting of even mild proximal aortic dilation.

One potential alternative to treat the disease of both the distal aorta and the iliac arteries is the use of unibody stent-grafts. The AFX (Endologix) stent-graft is a unibody, low-profile endograft aimed to treat abdominal aortic aneurysms. The particular configuration of this device and its so-called anatomical fixation make it potentially an optimal solution to overcome the issue reported before inherent to AIOD treatment. This device presents a unique design with its long main body and two innate limbs and is designed to be deployed and sits on the native aortoiliac bifurcation and represents the only one-piece bifurcated endograft designed to use anatomical fixation for endograft stabilization. The AFX device consists of a main bifurcated body and a proximal aortic extension, which fix firmly to the aorta and provides sealing while reducing the possibility of stent's migration at the same time. The skeleton of the device is made of a cobalt-chromium alloy in a multilinked self-expanding unibody. External to the stent, the fabric is made of multilayer ePTFE material (STRATA). The stent is attached only to the proximal and distal ends at the proximal aortic extension and allows ePTFE to move independently and conform to abnormal surfaces, facilitating the sealing of the sac. According to published literature, the unibody device seems to represent a valid choice in the treatment of abdominal aortic aneurysms, but this particular device would seem to satisfactorily perform even in the treatment of occlusive pathologies and recently has become part of our clinical practice.

Theoretical advantages of AFX (Endologix) are:

* Unibody design preserves aortic bifurcation, thanks to its anatomical fixation, as described previously. Unlike kissing stents (covered or uncovered), which can often protrude into the native aorta, disrupting flow and functionally raising the aortic bifurcation, a unibody device sits on and preserves the native bifurcation. This makes future "up-and-over" interventions to the lower extremities less technically challenging. Compared to CERAB, by using fewer stents in the narrow aorta, this technique has the added advantage of minimizing potential flow disturbances introduced by multiple covered stents.
* Graft fabric reduces neointimal hyperplasia: there is some evidence, including the randomized COBEST trial, that covered stents may be less likely to restenose or occlude than bare metal stents, particularly in TASC C and D lesions. This may be because the graft fabric represents a direct barrier to tissue ingrowth from neo-intimal hyperplasia.
* No limb competition in narrow bifurcation, thanks to its unibody design.
* Unibody stent-graft is protective in cases of potential ruptures, such as in heavily calcified lesions.
* Coverage of the entire diseased aorta may reduce atheroembolic risk. Using this covered graft and positioning it proximal and distal to the limits of disease effectively traps atherosclerotic material that could potentially embolize during device deployment, reducing atheroembolic risk.

As with any new treatment alternative, this treatment strategy has limitations.

* Compared with the placement of kissing stents, or even the CERAB technique, the AFX (Endologix) device requires a larger profile sheath (17-Fr ipsilateral sheath, 9-Fr contralateral).
* Placing a stent-graft also has a higher potential for coverage of collateral vessels.
* The procedure is more time-consuming and requires a higher level of endovascular technical skill.
* Finally, while cost-effectiveness cannot be evaluated without robust efficacy data and will fluctuate based upon local differences in costs, use of the AFX (Endologix) unibody stent-graft is likely to be more expensive than kissing stent placement.

The aim of the study is to evaluate the patency rates, safety, and efficacy of the AFX unibody stent-graft for the treatment of aortoiliac occlusive disease (AIOD), which may represent an additional technique in the endovascular treatment of this disease.

The results will demonstrate whether the AFX (Endologix) stent graft is effective for the treatment of AIOD, in particular in more complex lesions (TASC C and D). The effectiveness will be evaluated in terms of patency (primary, assisted and secondary), technical success, clinical success, and quality of life improvement. Other objectives are the evaluation of procedure-related adverse events and re-interventions, as well as operative details.

Nowadays, kissing stenting (KS) technique and the CERAB technique are considered the standard of care in the endovascular treatment of AIOD. However, patency rates and clinical success of the endovascular treatment, especially in the mid- and long- term, are still lower than the classic aorto-femoral bypass. Many aspects like the preservation of the aortic bifurcation, neointimal hyperplasia, limb competition, potential rupture, and atheroembolic risk are challenging problems that the endovascular surgeon has to face to improve the outcomes of the endovascular treatment. In vitro studies have investigated hemodynamic aspects15 but only three other groups have previously discussed their experience with this technique showing encouraging early- and mid-term results.

Compared to other endovascular procedures, AFX (Endologix) unibody endograft shows many risks and disadvantages:

* It is a more invasive procedure with a larger introducer (19F+7F), which may need a surgical access
* The cost of the procedure is higher if compared to KS (but similar to CERAB)
* The endograft has a risk of fabric laceration with high calcium volume
* Very low chronic outward force (COF) of the Elgiloy stent

ELIGIBILITY:
Inclusion Criteria:

* Age >18;
* Both sex;
* Preoperative 2.5mm CTA available;
* Written informed consent;
* Patients affected by AIOD classified as TASC B (with aortic involvement) C or D involving aortic bifurcation and or the first 5mm of one of both common iliacs;
* Treated in the coordinator center or in one of the study's participating center's;
* With a calcium volume in target zone based on real lumen of less than 20% and absence of circumferential calcifications;
* Minimum follow-up requested: 3-months, 12-18 months and 5-years CTA; clinical and DUS examination at 6- and 12- and 36-months after the intervention and yearly thereafter.

Exclusion Criteria:

* Age<18;
* No preoperative 2.5mm CTA available;
* Refused to sign the informed consent;
* Treated outside the coordinator centers or in one of the study's participating centers;
* Refusal to adhere to the requested follow-up;
* Patients affected by AIOD classified as TASC A or not involving aortic bifurcation or the first 5mm of one of both common iliacs;
* With a calcium volume in target zone based on real lumen of more than 20% and presence of circumferential calcifications;

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients affected by AIOD classified as TASC B, C or D involving aortic bifurcation and or the first 5mm of one of both common iliacs with indication to endovascular treatment enrolled at the Unit of Vascular Surgery of the Ospedale Civile di Baggiovara (Azienda Ospedaliero-Universitaria di Modena) and fulfilling the previous inclusion criteria. The Investigators (3 experts Vascular surgeons) will screen the patients for inclusion. Once the patient's eligibility will be stated, informed consent will be collected and the study could take place.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02-10 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Patency rate | through study completion, an average of 30 days (short), 1-year (mid) and 5-years (long)".
  short-, mid- and long-term patency rate (primary, assisted and secondary). Primary patency was defined as uninterrupted flow in the treated aortoiliac segment without occlusion or reintervention. Primary-assisted patency was defined as uninterrupted flow in the treated segment, allowing for reintervention for hemodynamically significant lesions in order to prevent occlusion. Secondary patency was defined as patency of the treated allowing for reintervention for occlusion.

SECONDARY OUTCOMES:
Technical success | within 24 hours of procedure conclusion
  Technical success, defined as insertion of the endograft with flow into both iliac arteries at the conclusion of the procedure.
Clinical Success | through study completion, an average of 30 days (short), 1-year (mid) and 5-years (long)".
  clinical success was defined as freedom from device-related death, conversion to open repair and graft limb thrombosis
Freedom from procedure related re-intervention and Adverse events | through study completion, an average 2-years.
  Adverse events are defined as any systemic or local complication directly related to the procedure. Adverse events that occurred in the first 30-day were considered procedure-related, unless differently demonstrated. Re-intervention were defined as any open surgical or endovascular procedure performed two correct an adverse events related to the procedure and/or device
Quality of life change | through study completion, an average 2-years.
  Improvement of quality of life will be measured as improvement of claudication interval
Rutherford scale change | through study completion, an average 2-years.
  Rutherford scale measures the severity of peripheral artery disease from a range of category between 0 (asymptomatic) to 6 (severe gangrene)
Cange of Ankle Brachial Index | through study completion, an average 2-years.
  Ankle Brachial Index (ABI) measures the ratio to the pressure at the anke and at the arm. It measures the grade of lower limb ischemia and range from 1.2 (normal) to 0 (critical ischemia).
Risk factor analysis | through study completion, an average of 30 days (short), 1-year (mid) and 5-years (long)".
  Analysis of anatomical and preoperative factors afflicting the primary outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- AOU di Modena, Baggiovara, Modena, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Maldonado TS, Westin GG, Jazaeri O, Mewissen M, Reijnen MM, Dwivedi AJ, Garrett HE Jr, Dias Perera A, Shimshak T, Mantese V, Smolock CJ, Arthurs ZM. Treatment of Aortoiliac Occlusive Disease with the Endologix AFX Unibody Endograft. Eur J Vasc Endovasc Surg. 2016 Jul;52(1):64-74. doi: 10.1016/j.ejvs.2016.04.003. Epub 2016 May 6. PMID 27162000
- [Background] Upchurch GR, Dimick JB, Wainess RM, Eliason JL, Henke PK, Cowan JA, Eagleton MJ, Srivastava SD, Stanley JC. Diffusion of new technology in health care: the case of aorto-iliac occlusive disease. Surgery. 2004 Oct;136(4):812-8. doi: 10.1016/j.surg.2004.06.019. PMID 15467666
- [Background] Aboyans V, Ricco JB, Bartelink MEL, Bjorck M, Brodmann M, Cohnert T, Collet JP, Czerny M, De Carlo M, Debus S, Espinola-Klein C, Kahan T, Kownator S, Mazzolai L, Naylor AR, Roffi M, Rother J, Sprynger M, Tendera M, Tepe G, Venermo M, Vlachopoulos C, Desormais I; ESC Scientific Document Group. 2017 ESC Guidelines on the Diagnosis and Treatment of Peripheral Arterial Diseases, in collaboration with the European Society for Vascular Surgery (ESVS): Document covering atherosclerotic disease of extracranial carotid and vertebral, mesenteric, renal, upper and lower extremity arteriesEndorsed by: the European Stroke Organization (ESO)The Task Force for the Diagnosis and Treatment of Peripheral Arterial Diseases of the European Society of Cardiology (ESC) and of the European Society for Vascular Surgery (ESVS). Eur Heart J. 2018 Mar 1;39(9):763-816. doi: 10.1093/eurheartj/ehx095. No abstract available. PMID 28886620
- [Background] Norgren L, Hiatt WR, Dormandy JA, Nehler MR, Harris KA, Fowkes FG; TASC II Working Group; Bell K, Caporusso J, Durand-Zaleski I, Komori K, Lammer J, Liapis C, Novo S, Razavi M, Robbs J, Schaper N, Shigematsu H, Sapoval M, White C, White J, Clement D, Creager M, Jaff M, Mohler E 3rd, Rutherford RB, Sheehan P, Sillesen H, Rosenfield K. Inter-Society Consensus for the Management of Peripheral Arterial Disease (TASC II). Eur J Vasc Endovasc Surg. 2007;33 Suppl 1:S1-75. doi: 10.1016/j.ejvs.2006.09.024. Epub 2006 Nov 29. No abstract available. PMID 17140820
- [Background] Grimme FA, Goverde PA, Van Oostayen JA, Zeebregts CJ, Reijnen MM. Covered stents for aortoiliac reconstruction of chronic occlusive lesions. J Cardiovasc Surg (Torino). 2012 Jun;53(3):279-89. PMID 22695260
- [Background] Sharafuddin MJ, Hoballah JJ, Kresowik TF, Sharp WJ, Golzarian J, Sun S, Corson JD. Long-term outcome following stent reconstruction of the aortic bifurcation and the role of geometric determinants. Ann Vasc Surg. 2008 May-Jun;22(3):346-57. doi: 10.1016/j.avsg.2007.12.013. Epub 2008 Apr 14. PMID 18411026
- [Background] Sabri SS, Choudhri A, Orgera G, Arslan B, Turba UC, Harthun NL, Hagspiel KD, Matsumoto AH, Angle JF. Outcomes of covered kissing stent placement compared with bare metal stent placement in the treatment of atherosclerotic occlusive disease at the aortic bifurcation. J Vasc Interv Radiol. 2010 Jul;21(7):995-1003. doi: 10.1016/j.jvir.2010.02.032. Epub 2010 Jun 11. PMID 20538478
- [Background] Mwipatayi BP, Thomas S, Wong J, Temple SE, Vijayan V, Jackson M, Burrows SA; Covered Versus Balloon Expandable Stent Trial (COBEST) Co-investigators. A comparison of covered vs bare expandable stents for the treatment of aortoiliac occlusive disease. J Vasc Surg. 2011 Dec;54(6):1561-70. doi: 10.1016/j.jvs.2011.06.097. Epub 2011 Sep 9. PMID 21906903
- [Background] Saratzis A, Salem M, Sabbagh C, Abisi S, Huasen B, Egun A, Nash J, Lau PF, Chaudhuri A, Dey R, Patrone L, Malina M, Davies R, Zayed H. Treatment of Aortoiliac Occlusive Disease With the Covered Endovascular Reconstruction of the Aortic Bifurcation (CERAB) Technique: Results of a UK Multicenter Study. J Endovasc Ther. 2021 Oct;28(5):737-745. doi: 10.1177/15266028211025028. Epub 2021 Jun 23. PMID 34160321
- [Background] Goverde PC, Grimme FA, Verbruggen PJ, Reijnen MM. Covered endovascular reconstruction of aortic bifurcation (CERAB) technique: a new approach in treating extensive aortoiliac occlusive disease. J Cardiovasc Surg (Torino). 2013 Jun;54(3):383-7. PMID 23640357
- [Background] Reijnen MM. Update on covered endovascular reconstruction of the aortic bifurcation. Vascular. 2020 Jun;28(3):225-232. doi: 10.1177/1708538119896197. Epub 2020 Jan 2. PMID 31896301
- [Background] Sirignano P, Silingardi R, Mansour W, Andreoli F, Migliari M, Speziale F. Unibody bifurcated aortic endograft: device description, review of the literature and future perspectives. Future Cardiol. 2021 Aug;17(5):793-804. doi: 10.2217/fca-2020-0119. Epub 2020 Nov 23. PMID 33225733
- [Background] Silingardi R, Sirignano P, Andreoli F, Mansour W, Migliari M, Speziale F; LIVE Study Collaborators. Unibody Endograft Using AFX 2 for Less Invasive and Faster Endovascular Aortic Repair: Protocol for a Multicenter Nonrandomized Study. JMIR Res Protoc. 2020 Apr 6;9(4):e16959. doi: 10.2196/16959. PMID 32250278
- [Background] Kouvelos GN, Nana P, Bouris V, Peroulis M, Drakou A, Rousas N, Giannoukas A, Matsagkas MI. Initial Clinical Experience with the Endologix AFX Unibody Stent Graft System for Treating Patients with Abdominal Aortic Aneurysms: A Case Controlled Comparative Study. Vasc Specialist Int. 2017 Mar;33(1):16-21. doi: 10.5758/vsi.2017.33.1.16. Epub 2017 Mar 31. PMID 28377907
- [Background] Chong A, Mirgolbabaee H, Sun Z, van de Velde L, Jansen S, Doyle B, Versluis M, Reijnen MMPJ, Groot Jebbink E. Hemodynamic Comparison of Stent-Grafts for the Treatment of Aortoiliac Occlusive Disease. J Endovasc Ther. 2021 Aug;28(4):623-635. doi: 10.1177/15266028211016431. Epub 2021 Jun 2. PMID 34076554
- [Background] Van Haren RM, Goldstein LJ, Velazquez OC, Karmacharya J, Bornak A. Endovascular treatment of TransAtlantic Inter-Society Consensus D aortoiliac occlusive disease using unibody bifurcated endografts. J Vasc Surg. 2017 Feb;65(2):398-405. doi: 10.1016/j.jvs.2016.08.084. Epub 2016 Oct 17. PMID 27765483
- [Background] Arnold A, Delaney CL, Wong YT, Wise N, Puckridge PJ. Reconstruction of the aorto-iliac segment in occlusive disease using the AFX unibody graft. ANZ J Surg. 2020 Dec;90(12):2496-2501. doi: 10.1111/ans.16236. Epub 2020 Aug 23. PMID 32830429
- [Background] Georgakarakos E, Ioannidis G, Koutsoumpelis A, Papatheodorou N, Argyriou C, Spanos K, Giannoukas AD, Georgiadis GS. Tauhe AFX unibody bifurcated unibody aortic endograft for the treatment of abdominal aortic aneurysms: current evidence and future perspectives. Expert Rev Med Devices. 2020 Jan;17(1):5-15. doi: 10.1080/17434440.2020.1704254. Epub 2019 Dec 20. PMID 31833437
- [Background] Rutherford RB, Baker JD, Ernst C, Johnston KW, Porter JM, Ahn S, Jones DN. Recommended standards for reports dealing with lower extremity ischemia: revised version. J Vasc Surg. 1997 Sep;26(3):517-38. doi: 10.1016/s0741-5214(97)70045-4. PMID 9308598

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-10): https://cdn.clinicaltrials.gov/large-docs/56/NCT05614856/Prot_SAP_000.pdf